CLINICAL TRIAL: NCT06415266
Title: Multicentric Randomized Study eValuating the sExual Quality of Life in Breast Cancer Patients Receiving oncoSexology Supportive Care on Proactive Versus On-request
Brief Title: Assessment the sExual Quality of Life in Breast Cancer Patients Receiving oncoSexology Supportive Care on Proactive Versus On-request
Acronym: VENUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2023-07 VEN; 2023-A02474-41 (Other: IDRCB)
Record Dates: First submitted 2024-04-17; First posted 2024-05-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: quality of sexual life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving oncoSexology supportive care on proactive (Experimental): Repeated assessment of the patient's needs in the field of oncosexology. Proposal of a personalized care plan to meet the various needs identified.
  Interventions: Other: Quality of life questionnaire (QLQ); Other: Satisfaction survey; Other: Assessment of patient needs in the field of oncosexology
- Patients receiving oncoSexology supportive care on request (Other): One-off distribution of a flyer to the patient containing both general information on sexual health and contact telephone numbers and e-mail addresses for oncosexology help
  Interventions: Other: Quality of life questionnaire (QLQ); Other: Satisfaction survey

INTERVENTIONS:
Other: Quality of life questionnaire (QLQ) — Quality of life questionnaire : EORTC QLQ-C30, EORTC QLQ-Breast cancer module (BR) 23, EORTC SHQ-C22 et HADS at inclusion, visit 1 (6 months +/-1 month before the inclusion), visit 2 (12 months +/-1 month before the inclusion), visit 3 (18 months +/-1 month before the inclusion) and visit 4 (24 months +/-1 month before the inclusion).
Other: Satisfaction survey — The satisfaction score will be collected using a visual analog scale from 0 to 10 and the satisfaction questionnaire will also be completed at visit 4 (24 months +/- 1 month before the inclusion).
Other: Assessment of patient needs in the field of oncosexology — Assessment of patient needs in the field of oncosexology during a face-to-face or virtual interview at inclusion and every 6 months for 2 years. If a need is identified, an oncosexology consultation will be organised. Following this, a personalised care plan may be proposed.
  Arms: Patients receiving oncoSexology supportive care on proactive

SUMMARY:
The study compares the quality of sexual life of breast cancer patients under two types of oncoSexology supportive care : personalized supportive care versus on-request. The aim is to improve the quality of sexual life of these patients.

DETAILED DESCRIPTION:
Breast cancer and its treatment are responsible for symptoms that can persist over time and affect quality of life. Given the improved prognosis for breast cancer, more and more patients are faced with the specific problems of the post-cancer period, and caring for them has become a major health issue. Sexual health is a crucial component of well-being and overall quality of life.

The study compares the quality of sexual life of breast cancer patients under two types of oncoSexology supportive care : personalized supportive care versus on-request.

For that, quality of life questionnaires will be completed by patients at inclusion and every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man at least 18 years old
* Diagnosis of infiltrating breast cancer regardless of the biological characteristics of the tumor
* Standard treatment by surgery, radiotherapy and/or chemotherapy, completed a maximum of 3 months ago with the exception of post-neoadjuvant treatments (chemotherapy, poly(ADP-ribose) polymerase (PARP) inhibitor, immunotherapy, targeted treatment, ...) which must have been started less than 3 months previously
* Patient with sufficient command of the French language to be able to answer the questionnaires
* Patient having given informed, written and express consent.
* Affiliation to the French Social Security System
* Willingness and ability to comply with scheduled visits, treatment plan and other study procedures

Exclusion Criteria:

* Patient already taken cared of in oncosexology. The following are not criteria for non-inclusion (a previous single consultation without treatment, use of local vaginal treatments)
* Metastatic disease
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of the quality of sexual life of patients in the intervention arm and patients in the control arm | at 12 months after the inclusion
  EORTC Sexual Health Questionnaire (SHQ)-C22 specific questionnaire sexual satisfaction scale score.
  Questionnaire comprising 2 multi-item scales assessing sexual satisfaction and dyspareunia; as well as 11 single items (including: importance of sexual activity, libido, incontinence, fatigue, impact of treatment on sexual life, communication with professionals, partner); as well as 4 items related to gender: 2 specific items for women (body image, vaginal dryness); 2 specific items for men (body image, confidence in maintaining an erection). The score ranges from 0 to 100. A high scale score represents a higher response level.

SECONDARY OUTCOMES:
Description of evolution in sexual quality of life | at inclusion, 6,12,18, and 24 months before inclusion
  Scores obtained on the EORTC SHQ-C22 questionnaire scales. Questionnaire comprising 2 multi-item scales assessing sexual satisfaction and dyspareunia; as well as 11 single items (including: importance of sexual activity, libido, incontinence, fatigue, impact of treatment on sexual life, communication with professionals, partner); as well as 4 items related to gender: 2 specific items for women (body image, vaginal dryness); 2 specific items for men (body image, confidence in maintaining an erection). The score ranges from 0 to 100. A high scale score represents a higher response level.
Description of evolution in quality of life - QLQ-C30 | at inclusion, 6,12,18, and 24 months before inclusion
  Scores obtained on the scales of the EORTC QLQ-C30. Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Description of evolution in quality of life - QLQ-Breast (BR)cancer module 23 questionnaires. | at inclusion, 6,12,18, and 24 months before inclusion
  Scores obtained on the scales of the QLQ-BR23 This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms.
Search for associations between comorbidities and risk factors | at inclusion, 6,12,18, and 24 months before inclusion
  Coefficients obtained with a model adapted for longitudinal quality of life data scores as a function of covariates potentially associated with sexual and global quality of life.
Search for associations between comorbidities and risk factors -questionnaire | at inclusion, 6,12,18, and 24 months before inclusion
  Anxiety and depression (psychological distress variables) will be assessed using the Hospital Anxiety and Depression Scale (HADS) questionnaire.
  The HADS is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a depression score (HADS-D), or can be added to produce a total score corresponding to emotional distress (HADS-T). Each item is rated on a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), for a total score ranging from 0-21 for each subscale. The entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Assessment of adherence to the programme in the interventional arm | at inclusion
  Percentage of adherence in the interventional arm
Oncosexology programme satisfaction | at 24 months before inclusion
  Satisfaction score measured on a visual analogue scale ranging from 1 to 10 (10 indicating high satisfaction)
Oncosexology programme satisfaction | at 24 months before inclusion
  Scores obtained of the Satisfaction questionnaire by arm. All the scale ranging from 1 to 5 (5 indicating high satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Véronique D'HONDT, Dr, Principal Investigator — Institut du Cancer de Montpellier (ICM)
Locations (9):
- France (9):
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Saint Herblain
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Vandoeuvre LES Nancy
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Institut Curie, Paris
  - IUCT - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Background] Carter J, Lacchetti C, Andersen BL, Barton DL, Bolte S, Damast S, Diefenbach MA, DuHamel K, Florendo J, Ganz PA, Goldfarb S, Hallmeyer S, Kushner DM, Rowland JH. Interventions to Address Sexual Problems in People With Cancer: American Society of Clinical Oncology Clinical Practice Guideline Adaptation of Cancer Care Ontario Guideline. J Clin Oncol. 2018 Feb 10;36(5):492-511. doi: 10.1200/JCO.2017.75.8995. Epub 2017 Dec 11. PMID 29227723
- [Background] Bobrie A, Jarlier M, Moussion A, Jacot W, D'Hondt V. Sexual quality of life assessment in young women with breast cancer during adjuvant endocrine therapy and patient-reported supportive measures. Support Care Cancer. 2022 Apr;30(4):3633-3641. doi: 10.1007/s00520-022-06810-3. Epub 2022 Jan 14. PMID 35028721
- [Background] Del Pup L, Villa P, Amar ID, Bottoni C, Scambia G. Approach to sexual dysfunction in women with cancer. Int J Gynecol Cancer. 2019 Mar;29(3):630-634. doi: 10.1136/ijgc-2018-000096. Epub 2019 Feb 13. PMID 30765487
- [Background] Dizon DS. Quality of life after breast cancer: survivorship and sexuality. Breast J. 2009 Sep-Oct;15(5):500-4. doi: 10.1111/j.1524-4741.2009.00766.x. Epub 2009 Jul 14. PMID 19614908
- [Background] Seguin L, Touzani R, Bouhnik AD, Charif AB, Marino P, Bendiane MK, Goncalves A, Gravis G, Mancini J. Deterioration of Sexual Health in Cancer Survivors Five Years after Diagnosis: Data from the French National Prospective VICAN Survey. Cancers (Basel). 2020 Nov 20;12(11):3453. doi: 10.3390/cancers12113453. PMID 33233583